CLINICAL TRIAL: NCT05665257
Title: Preoperative Inspiratory Muscle Training for Patients Undergoing Cytoreductive Surgery and Hyperthermic Intraperitoneal Chemotherapy - a Feasibility Study
Brief Title: Feasibility of Preoperative Inspiratory Muscle Training for Patients With Peritoneal Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ethical approval no 2016/338
Record Dates: First submitted 2022-12-05; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Peritoneal Metastases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training (Experimental): Participants in the intervention group were using a handheld device, Powerbreathe K3, aiming at increasing inspiratory muscle strength by applying an inspiratory resistance. They were instructed to use it twice a day for at least 14 days. Starting load was based on the baseline assessment of the participant's inspiratory muscle strength and increased during the intervention period.
  Interventions: Device: Inspiratory muscle training
- Mini-PEP (Sham Comparator): Participants in the control arm were instructed to use a handheld PEP-device traditionally used to facilitate deep breathing. The PEP-device does not provide any inspiratory resistance and therefore, it was considered a sham treatment. The control group were also instructed to use the device twice a day for at least two weeks.
  Interventions: Device: Mini-PEP

INTERVENTIONS:
Device: Inspiratory muscle training
  Arms: Inspiratory muscle training
Device: Mini-PEP
  Arms: Mini-PEP

SUMMARY:
The goal of this randomized controlled feasibility study was to evaluate the feasibility of preoperative inspiratory muscle training in patients undergoing surgery because of peritoneal metastases.

The main questions it aimed to answer was how feasible the intervention is regarding process and scientific feasibility as defined by Thabane et al 2010.

Participants in the intervention group were using a handheld device to increase their inspiratory muscle strength prior to surgery and researchers compared this group to a control group who were offered a sham treatment.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for cytoreductive surgery and hyperthermic intraperitoneal chemotherapy

Exclusion Criteria:

* Surgery scheduled less than two weeks from the date of inclusion
* Inability to speak and understand Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of preoperative inspiratory muscle training | The different outcome measures are assessed continuously during a period from inclusion until discharge from the hospital. This period varied in length (3 weeks-3 months) depending on when participants were scheduled for surgery.
  Feasibility will be assessed using two domains: process and scientific feasibility. These domains include several parts such as recruitment rates, time available for training, intervention adherence, patient acceptability, pre-and postoperative respiratory muscle and lung function assessments, reproducibility of assessments, preliminary treatment effect, incidence of PPCs, and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Andersson, PhD, Principal Investigator — Department of Medical Sciences, Respiratory, Allergy and Sleep Research, Uppsala University

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon reasonable request.